CLINICAL TRIAL: NCT02672267
Title: A Phase III, Double-blinded, Single Center, Randomized, Placebo Controlled Study to Assess the Safety, Tolerability, and Preliminary Efficacy of Single Intravenous Dose of Allogeneic Ischemia Tolerant Human Mesenchymal Bone Marrow Cells to Subjects With Acute Myocardial Infarction
Brief Title: A Study of Allogeneic Low Oxygen Mesenchymal Bone Marrow Cells in Subjects With Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Altaco XXI, LLP (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARDIO 1/2
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-04

CONDITIONS: Myocardial Infarction
Keywords: AMI, hBMMSCs, stem cells,
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cells (Experimental): Experimental: Stem Cells ALLOGENEIC LOW OXYGEN MESENCHYMAL BONE MARROW CELLS Intervention: Biological: Stem cells
  Interventions: Biological: Stem cells
- Placebo (Placebo Comparator): Lactated Ringer's Solution
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Stem cells — human Allogeneic Low Oxygen mesenchymal stem cells; Ischemia tolerant
  Other Names: Allogeneic Low Oxygen mesenchymal stem cells
  Arms: Stem Cells
Other: Placebo — Lactated Ringer's Solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and preliminary efficacy of human allogeneic ischemia tolerant mesenchymal bone marrow cells (aLoOxMBMC) administered intravenously to subjects with Acute Myocardial Infarction (STEMI, non STEMI).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains a leading cause of morbidity and mortality despite continuing advances in various treatment options. In developed countries, ischemic heart disease causes more than 50% of all cardiovascular deaths.

Stem cell transplantation has the potential to repair and improve cardiac function, thus helping to significantly decrease morbidity and mortality rates. Preclinical data from a variety of animal studies demonstrated the capacity for skeletal myoblasts to engraft, form myotubules, and enhance cardiac function after transplantation into infarcted myocardium. The underlying sequela of the post infarcted left ventricle often includes massive damage to the cardiomyocyte. The left ventricle remodeling (dilation) and dysfunction is thought to be irreversible. The development of treatments that will regenerate its musculature and vascular components is now considered a main therapeutic challenge. Preliminary human studies focusing on subjects with ischemic heart disease have demonstrated successful myoblast transplantation into the post infarction scar. Another study demonstrated the benefits of stem cell therapy on ventricular function and profusion.

Allogeneic mesenchymal stem cells have been used in a number of clinical trials for different indications. These clinical trials showed excellent safety, reduction in arrhythmias, improvement in functional status and increased ejection fraction.

The hMSCs are able to:

1. Prevent reperfusion injury;
2. Prevent excessive fibrosis;
3. Reestablish function of hibernating cardiomyocytes in peripheral zone area.
4. Reestablish angiogenesis/vasculogenesis;
5. Preserve wall motion (prevent arrhythmia and functional contractile deterioration);
6. Prevent post infarct ventricular remodeling and left ventricular dilation. It is well accepted that dilated cardiomyopathy mortality rates are 50% within 5 years of diagnosis;
7. Limit infarct size. If we can preserve and restore cardiac function as measured by ejection fraction and LVESV preserving left ventricular integrity would increase subject quality of life as well as longevity.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-85 years of age.
2. First Acute Myocardial Infarction (STEMI, non STEMI) within 7 days of study enrollment. Myocardial infarction is defined as ECG, Lab and CMR evidences.
3. Subject had successful revascularization within 12 hours of symptoms as evidenced by residual stenosis < 30% and TIMI antegrade flow II or III in the culprit vessel. Revascularization may include one of the following:

   * PCI angioplasty/stenting placement
   * Thrombolytic therapy
4. Life expectancy greater than 12 months.
5. Ability to understand and provide signed informed consent, or have a designated legal guardian or spouse legally able and willing to make such decisions on the subject's behalf.
6. Reasonable expectation that subject will receive standard post myocardial infarction care, unless contraindicated, including medications: • Anticoagulation (e.g. aspirin, clopidogrel, ticlopidine, prasugrel, etc.), beta-blockers, ace inhibitors, and statin agents, as tolerated.
7. Attend all scheduled safety follow-up visits.

Exclusion Criteria:

1. Hemodynamic instability as demonstrated by any of the following:

   * Requirement of intra-aortic balloon pump of left ventricular assist device.
   * Need for inotropic support (e.g. dopamine and/or dobutamine) for more than 36 hours for the maintenance of mean arterial blood pressure ≥60 mmHg.
2. History of cancer within the past 5 years, with the exception of localized basal or squamous cell carcinoma.
3. Clinically-significant hematologic, hepatic, or renal impairment within 24 hours of study procedure as determined by screening clinical laboratory tests. Severe chronic anemia or hematocrit ≤24%. Liver function tests (total bilirubin at 3 times upper limit of normal, or creatinine level ≥3mg/dL).
4. Presence of any other clinically-significant medical condition, psychiatric condition, or laboratory abnormality, that in the judgment of the Investigator or Sponsor for which participation in the study would pose a safety risk to the subject.
5. Participation in another study with an investigational drug or device within 3 months prior to stem cell administration.
6. History within the past year of drug or alcohol abuse.
7. Females known to be pregnant, lactating or having a positive pregnancy test (will be tested during screening) or planning to become pregnant during the study.
8. Inability to comply with the conditions of the protocol.
9. Presence of a transplanted tissue or organ or left ventricular assist device (LVAD) (or the expectation of the same within the next 12 months).
10. Planned Automatic Implantable Cardiac Defibrillator (AICD) or CRT within the next 12 months.
11. Need for chronic intermittent inotropic therapy.
12. Active myocarditis or early postpartum cardiomyopathy (within the first twelve months of delivery).
13. Porphyria.
14. Allergy to sodium citrate or any "caine" type of local anesthetic.
15. Subject scheduled for hospice care.
16. Clinically relevant abnormal findings in the clinical history, physical examination, ECG (e.g. life threatening arrhythmias, including QTc interval of ≥550 ms) or laboratory tests at the screening assessment that would interfere with the objectives of the study or that would, in the Investigator's opinion, preclude safe completion of the study.
17. Abnormal findings could include: known HIV infection or other immunodeficiency state, chronic active viral infection (such as hepatitis B or C), acute systemic infections (defined as subjects undergoing treatment with antibiotics), gastrointestinal tract bleeding, or any severe or acute concomitant illness or injury.
18. Any other medical, social, or geographical factor that would make it unlikely that the subject could comply with study procedures (e.g., alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location, or a history of noncompliance).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of aMBMC intravenous administration during the six month study period as determined by major adverse events MACE endpoint | 6 months

SECONDARY OUTCOMES:
The change from baseline on physical exam conducted at 1, 3 and 6 months post-administration | 6 months
LV end diastolic volume | 3 months
  measured by MRI
LV end systolic volume | 3 months
  measured by MRI
Infarct size measured by MRI, with contrast | 3 months
  measured by MRI
Global Left Ventricular Ejection Fraction | 3 months
  measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Saule Abseitova, MD, Prof., Principal Investigator — National Research Medical Center; Daniyar Jumaniyazov, MD, PhD, Study Director — Altaco XXI, LLP
Locations (1):
- National Research Medical Center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided